CLINICAL TRIAL: NCT03564626
Title: Health IT Generated PROs to Improve Outcomes in Cirrhosis
Acronym: HEROIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM20003950 multisite extension; 1R01HS025412-01A1 (AHRQ)
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard of care counseling and discharge instructions per local hospital policy. Standard of care follow up phone calls and visits at baseline and at 30 days. Follow-up will be for 30 days
- Health IT +/- Scheduled Follow Up (Experimental): Subjects and caregivers will be given individual phones loaded with the Patient Buddy App and the EncephalApp that will be used to enter medications, issues and orientation questions daily. There will be messages and phone calls as needed per the App and visits will be at baseline, scheduled at 15 days and at 30 days. In addition, scheduled phone calls will be performed at days 7 and 21.Follow-up will be for 30 days
  Interventions: Other: Health-IT +/- Scheduled Follow Up

INTERVENTIONS:
Other: Health-IT +/- Scheduled Follow Up — * Training patient and caregiver on Patient Buddy and EncephalApp
  * Counseling regarding readmission
  * Daily contact through app
  * Standard of care counseling regarding readmission and discharge instructions
  * Follow up phone calls at Week 1 and Week 3
  * In-person follow up visits at Week 2 and Week 4
  Arms: Health IT +/- Scheduled Follow Up

SUMMARY:
SPECIFIC AIM 1: To evaluate in a multi-center, randomized trial the effectiveness of PROs elicited using PatientBuddy and EncephalApp on the prevention of avoidable 30 day readmissions in patients with cirrhosis and their caregivers compared to standard of care.

DETAILED DESCRIPTION:
Cirrhosis affects more than 6 million US patients and is a major burden on patients, caregivers and the healthcare system. Patients with cirrhosis are prone to clinical and psycho-social issues that may predict hospitalization, re-hospitalizations and death. Important patient-reported outcomes (PRO) such as impaired daily functioning, sleep, cognition and pain are widely prevalent in patients with cirrhosis. These changes can independently impact hospitalizations, re-hospitalizations and death in cirrhotic patients. The investigators have studied the impact of these PRO using traditional and computerized scales such as PROMIS (Patient-reported outcomes measurement information system). With the increasing spread of health-related electronic devices, the relevance of health IT in the management of chronic diseases such as cirrhosis is paramount. The team has already developed and used several health IT advances to educate patients and their caregivers in inpatient and outpatient settings. These tools are Patient Buddy to define patients regarding factor preventing readmission, and EncephalApp Stroop to detect cognitive dysfunction in cirrhosis. As part of a funded AHRQ R21, PatientBuddy, which has undergone multiple refinements in response to feedback from patients, caregivers and administering staff, is being used by the study team to prevent readmissions to Virginia Commonwealth University Medical Center (VCU). However the evaluation of these tools in a multi-center study that adapts to the status of the patients and their caregivers is an important step towards improvement in cirrhosis-related outcomes. In addition, PROs that are elicited and monitored when the patients are outside the hospital will advance the field by making them integral parts of clinical management.

ELIGIBILITY:
Patient Inclusion Criteria:

* Cirrhosis patients ≥21 years of age hospitalized for non-elective reasons
* Adult caregiver and the patient living in the same house
* Able to complete the Patient Buddy training and evaluation
* Discharged home from the hospital
* Discharge hospital as primary hospital base

Caregiver Inclusion Criteria:

* Living in same dwelling as patient for the last ≥1 year
* Able to complete the Patient Buddy training and evaluation
* Familiar with the patient's routine

Patient Exclusion Criteria:

* Elective hospitalization
* Lack of an adult caregiver
* Active substance abuse within 1 month of the hospitalization (alcohol use is acceptable provided the patient does not have alcoholic hepatitis during this admission or <1 month prior to admission)
* Unable to perform training or give consent
* Patients discharged to hospice, nursing home or extended care facilities
* pregnant women
* patients with limited English proficiency

Caregiver Exclusion Criteria

* Unable or unwilling to train or adhere to study guidelines
* Unfamiliar with the patient routines
* Not in the same house as the patient

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — VCU Medical Center
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Acharya C, Sehrawat TS, McGuire DB, Shaw J, Fagan A, McGeorge S, Olofson A, White MB, Gavis E, Kamath PS, Bergstrom L, Bajaj JS. Perspectives of Inpatients With Cirrhosis and Caregivers on Using Health Information Technology: Cross-sectional Multicenter Study. J Med Internet Res. 2021 Apr 9;23(4):e24639. doi: 10.2196/24639. PMID 33744844

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group/Not Dyad: Standard of care counseling and discharge instructions per local hospital policy. Standard of care follow up phone calls and visits at baseline and at 30 days. Follow-up will be for 30 days. No dyads enrolled in this part of the study. Only the patients (subjects) were enrolled in this part of the study, not dyads. The numbers only represent the patient enrollment numbers.
- Health IT +/- Scheduled Follow Up/ no Dyads: No dyads enrolled. Subjects will be given individual phones loaded with the Patient Buddy App and the EncephalApp that will be used to enter medications, issues and orientation questions daily. There will be messages and phone calls as needed per the App and visits will be at baseline, scheduled at 15 days and at 30 days. In addition, scheduled phone calls will be performed at days 7 and 21.Follow-up will be for 30 days
  Health-IT +/- Scheduled Follow Up: -Training patient on Patient Buddy and EncephalApp
  * Counseling regarding readmission
  * Daily contact through app
  * Standard of care counseling regarding readmission and discharge instructions
  * Follow up phone calls at Week 1 and Week 3
  * In-person follow up visits at Week 2 and Week 4
Period: Overall Study
Arm/Group | Control Group/Not Dyad | Health IT +/- Scheduled Follow Up/ no Dyads
Started | 116 | 116
Completed | 116 | 116
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group/ no Dyads: Standard of care counseling and discharge instructions per local hospital policy. Standard of care follow up phone calls and visits at baseline and at 30 days. Follow-up will be for 30 days. No dyads enrolled in this part of the study. Only the patients (subjects) were enrolled in this part of the study, not dyads. The numbers only represent the patient enrollment numbers.
- Health IT +/- Scheduled Follow Up/ no Dyads: Subjects will be given individual phones loaded with the Patient Buddy App and the EncephalApp that will be used to enter medications, issues and orientation questions daily. There will be messages and phone calls as needed per the App and visits will be at baseline, scheduled at 15 days and at 30 days. In addition, scheduled phone calls will be performed at days 7 and 21.Follow-up will be for 30 days
  Health-IT +/- Scheduled Follow Up: -Training patient on Patient Buddy and EncephalApp
  * Counseling regarding readmission
  * Daily contact through app
  * Standard of care counseling regarding readmission and discharge instructions
  * Follow up phone calls at Week 1 and Week 3
  * In-person follow up visits at Week 2 and Week 4
- Total: Total of all reporting groups
Arm/Group | Control Group/ no Dyads | Health IT +/- Scheduled Follow Up/ no Dyads | Total
Number analyzed (Participants) | 116 | 116 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.42 (8.89) | 59.1 (12.38) | 58.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 58 | 98
  Male | 76 | 58 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 110 | 110 | 220
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 36 | 53 | 89
  White | 80 | 63 | 143
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 116 | 116 | 232

OUTCOME MEASURES:

1. Primary Outcome: Avoidable Readmissions
Description: Avoidable readmissions within 30 days
Time Frame: 30 days
Measure: Number; unit: Number of avoidable readmissions
Groups:
- Control Group/ No Dyads: Standard of care counseling and discharge instructions per local hospital policy. Standard of care follow up phone calls and visits at baseline and at 30 days. Follow-up will be for 30 days. Just the patients counted and reported, not the dyads.
Arm/Group | Control Group/ No Dyads | Health IT +/- Scheduled Follow Up/ no Dyads
Number analyzed (Participants) | 116 | 116
Number of avoidable readmissions | 12 | 23

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Control Group/ no Dyads: Standard of care counseling and discharge instructions per local hospital policy. Standard of care follow up phone calls and visits at baseline and at 30 days. Follow-up will be for 30 days. Only the subjects were counted, not the dyads.
- Health IT +/- Scheduled Follow Up/ no Dyads: Subjects (not dyads) will be given individual phones loaded with the Patient Buddy App and the EncephalApp that will be used to enter medications, issues and orientation questions daily. There will be messages and phone calls as needed per the App and visits will be at baseline, scheduled at 15 days and at 30 days. In addition, scheduled phone calls will be performed at days 7 and 21.Follow-up will be for 30 days
  Health-IT +/- Scheduled Follow Up: -Training patient on Patient Buddy and EncephalApp
  * Counseling regarding readmission
  * Daily contact through app
  * Standard of care counseling regarding readmission and discharge instructions
  * Follow up phone calls at Week 1 and Week 3
  * In-person follow up visits at Week 2 and Week 4
Arm/Group | Control Group/ no Dyads | Health IT +/- Scheduled Follow Up/ no Dyads
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/116
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/116
Other Adverse Events (participants affected / at risk) | 0/116 | 0/116

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03564626/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03564626/ICF_000.pdf